CLINICAL TRIAL: NCT06636006
Title: Effects of Aerobic Exercise Versus Digital Cognitive Behavioral Therapy for Insomnia in University Students with Insomnia Complaints
Brief Title: Aerobic Exercise Versus Digital Cognitive Behavioral Therapy for Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Associate professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI05992-2024
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-10

CONDITIONS: Insomnia Chronic
Keywords: chronic insomnia; exercise; sleep; anxiety; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity; Anxiety Disorders; Depression | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise (Experimental): Three sessions of aerobic exercise per week (outdoor walking), for 50 continuous minutes, at moderate intensity (Identified by the Borg Subjective Perception of Exertion Scale, scores from 12 to 13), will be performed for 7 weeks. These sessions will be accompanied by a researcher responsible for data collection, who will make a daily record of the activities. The practice time will be between 5:00 pm and 7:00 pm.
  Interventions: Behavioral: Aerobic Exercise
- Digital Cognitive Behavioral Therapy (CBT-I) (Active Comparator): Three weekly sessions of digital CBT-I will be held through the Vigilantes do Sono® application (digital therapy with the therapeutic protocol approved by ANVISA, Brazil).

INTERVENTIONS:
Behavioral: Aerobic Exercise — 50 continuous minutes, at moderate intensity (Identified by the Borg Subjective Perception of Exertion Scale, scores from 12 to 13)
  Arms: Aerobic Exercise
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I includes some therapies, including sleep restriction therapy, stimulus control therapy, sleep hygiene education, relaxation and cognitive therapy[19]. Traditionally, CBT-I is applied in person (individually or in a group) by a trained psychologist or psychiatrist. However, several studies show similar effects when CBT-I is performed remotely, and online (digital)

SUMMARY:
The purpose of this study is to compare the effects of aerobic exercise versus digital CBT-I in university students with insomnia complaints. This is a clinical trial. Participants will be randomized into two groups: aerobic exercise (n=25) and digital CBT-I (n=25). The severity of insomnia, sleep quality, pre-sleep cognitive and somatic arousal, and participants' complaints of depression, anxiety, and stress will be assessed using self-administered questionnaires. Based on previous studies describing the effects of physical exercise on chronic insomnia, the hypothesis of this study is that aerobic exercise promotes similar results compared to digital CBT-I in insomnia severity and sleep quality, in addition to improving the complaints of depression, anxiety and stress of the participants.

ELIGIBILITY:
Inclusion Criteria:

* ages ≥ 18 years old
* insomnia severity index score >8
* be physically inactive according to the IPAQ questionnaire

Exclusion criteria:

* non-adherence to intervention protocols
* absence or incomplete answers in the questionnaires/evaluation methods of the study
* shift workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | baseline and post-intervention (7 weeks)
  The severity of insomnia will be assessed using the Insomnia Severity Index (ISI) questionnaire. This instrument was developed to assess insomnia complaints. It is a self-administering, brief and simple scale, composed of 7 items that can be classified from 0 to 4, with the lowest final score = 0 and the highest = 28. Scores from 0 to 7 are considered non-significant insomnia, lower limit for insomnia from 8 to 14, moderate insomnia from 15 to 21, and severe insomnia from 22 to 28

SECONDARY OUTCOMES:
Physical evaluation and Anamnesis | baseline and post-intervention (7 weeks)
  To evaluate the changes in the body composition (body mass, % fat and fat-free mass) of participants, a bioimpedance scale (Omron, HBF-514) will be used, with a capacity of up to 150kg. Height will be assessed by stadiometer (Sanny, Professional). The Body Mass Index (body mass/height 2) will be calculated. An anamnesis form will be used to record the participants' personal information such as age, gender, use of medications, etc
Cognitive and somatic arousal | baseline and post-intervention (7 weeks)
  To assess the level of pre-sleep cognitive and somatic arousal, the self-reported questionnaire will be used Pre-Sleep Arousal Scale (PSAS), composed of 16 items, 8 of which assess cognitive alertness and 8 assess somatic alertness. Each item has a 5-point scale that determines the intensity of the symptom experienced at the onset of sleep, with a score of 1 being no symptoms experienced and a score of 5 expressing an extremely intense symptom.
Sleep Quality | baseline and post-intervention (7 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess the sleep quality over the past 30 days. An overall score of 5 or less indicates good sleep quality, whereas scores greater than 5 indicate poor sleep quality.
Sleep Diary | baseline and post-intervention (7 weeks)
  The sleep diary is a method used to assess the subjective perception of sleep quality, so it should be answered in the morning upon waking. The questions contained in this questionnaire are related to bedtime and wake-up times, the number of hours of sleep, latency to sleep onset, and awakenings during the night.
Symptoms of anxiety, depression, and stress | baseline and post-intervention (7 weeks)
  Depression Anxiety Stress Scale-21 (DASS-21) will be used to evaluate anxiety, depression and stress. It is an instrument composed of a self-report scale that contains a set of three subscales type Likert of four points 0, 1, 2 and 3, where zero (strongly disagree) and three (strongly agree). Each subscale of the DASS-21 It consists of seven items. The variations in the scores correspond to the severity of the symptoms for each subscale, which vary between "normal", "minimal", "mild", "moderate", "severe and "very severe". The scores of each subscale were calculated by summing the scores of the seven items, multiplied by two.
Physical activity level | baseline and post-intervention (7 weeks)
  The short version of the International Physical Activity Questionnaire (IPAQ-SF) will be used to assess the level of physical activity of the participants, with reference to the activities of the last week. The questionnaire consists of questions regarding the frequency and duration of moderate, vigorous, and walking physical activities. Participants will be classified as insufficiently active (<150 minutes of moderate activity/week) and active (≥150 minutes of moderate activity).
Sedentary Behavior | baseline and post-intervention (7 weeks)
  Sedentary behavior will be assessed using time spent sitting during a typical weekday and weekend. The following equation will be applied to calculate the average sitting time per day: [(week x 5) + (weekend x 2)] / 7. Daily sitting time classified into 3 categories (<8 hours per day, ≥ 8 to < 11 hours a day and ≥ 11 hours a day).

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Tereza, Jatai, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vignola RC, Tucci AM. Adaptation and validation of the depression, anxiety and stress scale (DASS) to Brazilian Portuguese. J Affect Disord. 2014 Feb;155:104-9. doi: 10.1016/j.jad.2013.10.031. Epub 2013 Oct 28. PMID 24238871
- [Background] Rosenberg DE, Bull FC, Marshall AL, Sallis JF, Bauman AE. Assessment of sedentary behavior with the International Physical Activity Questionnaire. J Phys Act Health. 2008;5 Suppl 1:S30-44. doi: 10.1123/jpah.5.s1.s30. PMID 18364524
- [Background] Matsudo, S., Araújo, T., Matsudo, V., Andrade, D., Andrade, E., Oliveira, L. C., Braggion, G. International Physical Activity Questionnaire (IPAQ): Validity and reproducibility study in Brazil. . Brazilian Journal of Physical Activity and Health. 2001,5:5-18.
- [Background] Ruivo Marques D, Allen Gomes A, Nicassio PM, Azevedo MHP. Pre-Sleep Arousal Scale (PSAS): psychometric study of a European Portuguese version. Sleep Med. 2018 Mar;43:60-65. doi: 10.1016/j.sleep.2017.10.014. Epub 2017 Dec 19. PMID 29482814
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786